CLINICAL TRIAL: NCT05847569
Title: Phase II Trial for Evaluation of Alternate Doses and Dosing Schedules of Belantamab Mafodotin in Triple-Class Refractory Multiple Myeloma
Brief Title: Alternate Doses and Dosing Schedules of Belantamab Mafodotin for Treatment of Triple-Class Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC210812; NCI-2023-03039 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC210812 (Other: Mayo Clinic); 22-001207 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; Specimen Handling; Fluid Therapy; Biopsy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (low dose belantamab mafodotin) (Active Comparator): Patients receive low dose belantamab mafodotin intravenously (IV) on day 1 of each cycle. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. All patients undergo a CT scan, a MRI scan, or a PET/CT scan during screening and patients with plasmacytoma (a MM tumor in bone or soft tissue) also undergo imaging scans on study. Patients undergo bone marrow aspirate and biopsy during screening and on study as well as collection of blood samples throughout the trial.
  Interventions: Biological: Belantamab Mafodotin; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography
- Group II (low dose and high dose belantamab mafodotin) (Experimental): Patients receive belantamab mafodotin IV on day 1. Cycle repeats at 3 weeks for the next cycle and then every 6 weeks for subsequent cycles in the absence of disease progression or unacceptable toxicity. All patients undergo a CT scan, a MRI scan, or a PET/CT scan during screening and patients with plasmacytoma (a MM tumor in bone or soft tissue) also undergo imaging scans on study. Patients undergo bone marrow aspirate and biopsy during screening and on study as well as collection of blood samples throughout the trial.
  Interventions: Biological: Belantamab Mafodotin; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Belantamab Mafodotin — Given IV
  Other Names: Belantamab Mafodotin-blmf; Blenrep; GSK2857916; J6M0-mcMMAF
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspirate — Undergo bone marrow aspirate
  Other Names: BONE MARROW, LIQUID; Human Bone Marrow Aspirate
Procedure: Bone Marrow Biopsy — Undergo biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography; Computerized Tomography (CT) scan
Procedure: Magnetic Resonance Imaging — Undergo MRI scan
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; Magnetic Resonance Imaging (MRI)
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial tests alternate doses and dosing schedules of belantamab mafodotin in treating patients with triple-class multiple myeloma that has come back (after a period of improvement) (recurrent) and/or does not respond to treatment (or that has not responded to previous treatment) (refractory). Belantamab mafodotin is a monoclonal antibody, belantamab, linked to a chemotherapy drug, mafodotin. Belantamab is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, known as BCMA receptors, and delivers mafodotin to kill them. This trial may help researchers determine if alternate doses and dosing schedules work better in preventing certain side effects, such as eye toxicity, and treating patients with recurrent or refractory multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the grade 3/4 keratopathy-free rate at the time of dose #4 of an alternative dose/dosing schedule of belantamab mafodotin in patients with relapsed or refractory multiple myeloma (RRMM).

SECONDARY OBJECTIVES:

I. To assess the overall response rate (ORR; partial response or better) of an alternative dose/dosing schedule of belantamab mafodotin in patients with RRMM.

II. To assess the safety of an alternative dose/dosing schedule of belantamab mafodotin in patients with RRMM.

III. To assess the time to progression (TTP) of an alternative dose/dosing schedule of belantamab mafodotin in patients with RRMM.

IV. To assess the progression free survival (PFS) with an alternative dose/dosing schedule of belantamab mafodotin in patients with RRMM.

V. To assess the overall survival (OS) with an alternative dose/dosing schedule of belantamab mafodotin in patients with RRMM.

VI. To assess the minimal residual disease (MRD) negativity rate in patients who have achieved a complete response (CR) with an alternative dose/dosing schedule of belantamab mafodotin.

CORRELATIVE AND PHARMACODYNAMIC RESEARCH OBJECTIVES:

I. To assess the association of pre-treatment serum BCMA levels as well as serum BCMA levels throughout treatment with ORR and PFS to an alternative treatment schedule of belantamab mafodotin.

II. To assess the pharmacokinetics of this alternative dose/dosing schedule of belantamab mafodotin.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive low dose belantamab mafodotin intravenously (IV) on day 1 of each cycle. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. All patients undergo a computed tomography (CT) scan, a magnetic resonance image (MRI) scan, or a positron emission tomography (PET)/CT scan during screening and patients with plasmacytoma (a multiple myeloma [MM] tumor in bone or soft tissue) also undergo imaging scans on study. Patients undergo bone marrow aspirate and biopsy during screening and on study as well as collection of blood samples throughout the trial.

GROUP II: Patients receive belantamab mafodotin IV on day 1. Cycle repeats at 3 weeks for the next cycle and then every 6 weeks for subsequent cycles in the absence of disease progression or unacceptable toxicity. All patients undergo a CT scan, a MRI scan, or a PET/CT scan during screening and patients with plasmacytoma (a MM tumor in bone or soft tissue) also undergo imaging scans on study. Patients undergo bone marrow aspirate and biopsy during screening and on study as well as collection of blood samples throughout the trial.

After completion of trial treatment, patients are followed up every 12 weeks for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, 2
* Histologically or cytologically confirmed diagnosis of multiple myeloma (MM), as defined in International Myeloma Working Group (IMWG) criteria, and:

  * If patients have undergone stem cell transplantation (SCT), day 0 of SCT must be > 100 days prior to registration to be eligible for the study
  * Has had disease progression after >= 3 prior lines of anti-myeloma treatments including one proteasome inhibitor (eg. bortezomib, carfilzomib or ixazomib), one immunomodulatory agent (eg.thalidomide, lenalidomide or pomalidomide) and one anti-CD38 monoclonal antibody (eg.daratumumab or isatuximab)
  * Prior non-belantamab mafodotin anti-BCMA agent exposure is allowed; patients with prior treatment with an anti-BCMA chimeric antigen receptor (CAR)-T or bispecific antibody will be allowed to participate in the study
* Has measurable disease with at least one of the following:

  * Serum M-protein >= 0.5 g/dL (>= 5 g/L)
  * Urine M-protein >= 200 mg/24 h
  * Serum free light chain (FLC) assay: Involved FLC level >= 10 mg/dL (>= 100 mg/L) and an abnormal serum free light chain ratio (< 0.26 or > 1.65)
  * Note: Patients with non-secretory disease will be allowed to participate
* Absolute neutrophil count >= 0.75 x 10^9/L (=< 28 days prior to registration)

  * Without growth factor support, blood transfusion, or platelet stimulating agents for the past 14 days, excluding erythropoietin
* Hemoglobin >= 7.0 g/dL (=< 28 days prior to registration)

  * Without growth factor support, blood transfusion, or platelet stimulating agents for the past 14 days, excluding erythropoietin
* Platelets >= 50 x 10^9/L (=< 28 days prior to registration)

  * Without growth factor support, blood transfusion, or platelet stimulating agents for the past 14 days, excluding erythropoietin
* Total bilirubin =< 2.0 x upper limit of normal (ULN) (=< 28 days prior to registration); (total bilirubin >= 2.0 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is < 35%)
* Alanine aminotransferase =< 2.5 x ULN (=< 28 days prior to registration)
* Aspartate transaminase =< 2.5 x ULN (=< 28 days prior to registration)
* Estimated glomerular filtration rate (eGFR) >= 30 mL/min/1.73 m^2 (=< 28 days prior to registration)

  * As calculated by Modification of Diet in Renal Disease (MDRD) formula
* Spot urine [albumin/creatinine ratios (spot urine)] =< 500 mg/g (56 mg/mmol) OR urine dipstick negative/trace [if >1+ only eligible if confirmed =< 500 mg/g (56 mg/mmol) by albumin/creatinine ratio (spot urine from first void)] (=< 28 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only. Both females and males must agree to follow the instructions

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Provide written informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the study protocol
* Willingness to provide mandatory blood specimens for correlative research
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

Exclusion Criteria:

* Active plasma cell leukemia at the time of screening. Symptomatic amyloidosis, active POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal plasmaproliferative disorder, myeloma protein, and skin changes), Waldenstrom Macroglobulinemia
* Prior belantamab mafodotin therapy. However, patients with prior exposure to another non-belantamab mafodotin anti-BCMA agent such as an anti-BCMA CAR-T or anti-BCMA bispecific antibody will be allowed to participate in the study
* Systemic active infection requiring treatment
* Any unresolved toxicity >= grade 2 from previous treatment except for alopecia, or peripheral neuropathy up to grade 2
* Any major surgery =< 4 weeks prior to registration
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities except renal impairment) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures
* Evidence of active mucosal or internal bleeding
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if participant otherwise meets entry criteria
* Participants with previous or concurrent malignancies other than multiple myeloma are excluded, unless the prior malignancy has been considered medically stable for > 2 years. The participant must not be receiving active therapy, other than hormonal therapy for this disease. NOTE: Participants with curatively treated nonmelanoma skin cancer are allowed without a 2-year restriction.
* Evidence of cardiovascular risk, including any of the following:

  * Evidence of current clinically significant untreated arrhythmias, including clinically significant electrocardiogram (ECG) abnormalities including 2nd degree (Mobitz type II) or 3rd degree atrioventricular (AV) block
  * History of myocardial infarction (=< 6 months), acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 12 weeks of screening
  * Class III or IV heart failure as defined by the New York Heart Association functional classification system [NYHA, 1994]
  * Uncontrolled hypertension
* Known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs chemically related to belantamab mafodotin, or any of the components of the study treatment
* Known human immunodeficiency virus (HIV) infection, unless the participant can meet all of the following criteria:

  * Established anti-retroviral therapy (ART) for at >=4 weeks and HIV viral load < 400 copies/mL
  * CD4+ T-cell (CD4+) counts >= 350 cells/uL
  * No history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections < 12 months prior
  * Note: consideration must be given to ART and prophylactic antimicrobials that may have a drug-drug interaction and/or overlapping toxicities with belantamab mafodotin or other combination products as relevant
* Patients with hepatitis B will be excluded unless the following criteria can be met:

  * If patient's serology shows hepatitis B virus core antibody (HbcAb)+ and hepatitis B surface antigen (HbsAg)-, they must have undetectable hepatitis B virus (HBV) deoxyribonucleic acid (DNA) at screening. Patients will be monitored per protocol. Antiviral treatment would be instituted if HBV DNA becomes detectable
  * If patient's serology shows HBsAg+ at screen or within 3 months prior, patients must have undetectable HBV DNA at screening, must have started highly effective antiviral treatment at least 4 weeks prior to registration, and must have baseline imaging per protocol (patients with cirrhosis are excluded). Patients must remain on antiviral treatment throughout the study. Patients will be monitored per protocol
  * Note: presence of hepatitis (Hep) B surface antibody (HBsAb) indicating previous vaccination will not exclude a participant.
* Positive hepatitis C antibody test result or positive hepatitis C ribonucleic acid (RNA) test result at screening or =< 12 weeks prior to first dose of study treatment unless the participant can meet the following criteria:

  * RNA test negative
  * Successful anti-viral treatment (usually 8 weeks duration) is required, followed by a negative HCV RNA test after a washout period >= 4 weeks
* Current corneal epithelial disease except for mild punctuate keratopathy
* Participant who received plasmapheresis within =< 7 days prior to registration
* Patients who received prior allogeneic stem cell transplant
* Participant who received a live or live-attenuated vaccine =< 30 days prior to registration. Ok to receive coronavirus disease (COVID) vaccine at any timepoint during protocol treatment
* Participant is a woman who is pregnant or lactating
* Participant who plans on wearing contact lenses during treatment with belantamab mafodotin

Lifestyle Considerations:

Contact lenses are prohibited for participants while they are receiving belantamab mafodotin treatment. Contact lens use may be restarted after belantamab mafodotin treatment is discontinued, provided a qualified eye care specialist confirm there are no other contraindications. Use of bandage contact lenses is allowed for the treatment of corneal epithelial disease as prescribed by an ophthalmologist/eye care professional.

No other lifestyle restrictions are required for participants in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2029-06-29 (Estimated); Study Completion 2034-06-29 (Estimated)

PRIMARY OUTCOMES:
Grade 3/4 keratopathy-free rate | At the time of dose 4
  The proportion of successes will be estimated by the number of successes (proportion of patients free of grade 3/4 keratopathy at the time of dose #4) divided by the total number of evaluable patients. 95% confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner. If both arms prove to meet the primary endpoint, they will be evaluated indirectly in relation to each other similar, to a Bayesian pick the winner, approach if only one can be brought forward for further testing

SECONDARY OUTCOMES:
Overall response rate | Up to 5 years
  Will be estimated by the total number of patients who achieve a complete response (CR), very good partial response, or partial response divided by the total number of evaluable patients. All evaluable patients will be used for this analysis. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Incidence of adverse events (AEs) | Up to 5 years
  The maximum grade for each type of AE will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the AEs to the study treatment will be taken into consideration.
Time to progression | From registration to the earliest date of documentation of disease progression, assessed up to 5 years
  The distribution of time will be estimated using the method of Kaplan-Meier.
Progression free survival (PFS) | From registration to the earliest date of documentation of disease progression or relapse or death due to any cause, assessed up to 5 years
  The distribution of PFS will be estimated using the method of Kaplan-Meier.
Overall survival (OS) | From registration to death due to any cause, assessed up to 5 years
  The distribution of OS will be estimated using the method of Kaplan-Meier.
Minimal residual disease (MRD) negativity rate | Up to 5 years
  Will be estimated by dividing the total number of patients who achieve MRD negativity if a bone marrow biopsy is done for suspected CR over the total number of evaluable patients. All evaluable patients will be used for this analysis. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo D. Parrondo, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials